CLINICAL TRIAL: NCT06448143
Title: An Open-Label, Multicenter Study to Evaluate the Safety, Pharmacokinetics and Conspicuity of Bludigo® When Used as an Aid in the Determination of Ureteral Patency in Pediatric Patients
Brief Title: Indigotindisulfonate Sodium Injection, USP as an Aid in the Determination of Ureteral Patency in Pediatric Patients
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Prove pharm (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PVP-21IC03
Record Dates: First submitted 2024-05-20; First posted 2024-06-07 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Ureter Injury
MeSH Terms: interventions — Indigo Carmine; Injections

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Weight-based dose (Experimental): open label evaulation of weight based dose of Bludigo
  Interventions: Drug: Indigotindisulfonate sodium 0.8% injection

INTERVENTIONS:
Drug: Indigotindisulfonate sodium 0.8% injection — Experimental contrast dye for diagnostic procedures, commonly used as a visualization aid in pelvic and abdominal surgeries, as well as for evaluating ureteral patency.
  Other Names: Bludigo®

SUMMARY:
This is an open-label, multicenter study to evaluate the safety, pharmacokinetics, and conspicuity of a weight-based Bludigo® dose (0.05 mL/kg rounded up (if necessary) to a minimum of 0.5 mL and not to exceed 2.5 mL) when used as an aid in the determination of ureteral patency in pediatric patients.

The study will enroll approximately 18 pediatric patients from approximately 2-3 study centers in the United States.

Patients scheduled for urological or gynecological surgical procedures who are < 17 years will be screened for participation.

A minimum of 6 patients will be enrolled in each of the following three age groups: birth to <6-years old, 6 to < 12 years old, 12 to < 17 years old.

Screening will occur within 30 days before study drug administration (Day of Surgery).

After signing the informed consent, review of inclusion and exclusion criteria will be performed. The collection of medical history and concomitant medications, the completion of a physical examination including vital signs measurement, ECG, and the collection of baseline laboratory testing (samples must be collected within 14 days of day 1) will be completed during the screening period.

On the Day of Surgery (Day 1) patients will be evaluated for eligibility for treatment.

To evaluate the efficacy outcomes, each patient will be injected with a weight-based dose of Bludigo® (0.05 mL/kg rounded up (if necessary) to a minimum of 0.5 mL) the maximum dose to be injected is not to exceed 2.5 mL. The ureteral orifices / urine jet will be observed, and a video will be recorded for 10 minutes. The time that will be captured on video is from the time of Bludigo® injection to 10 minutes post injection. If both ureters cannot be visualized simultaneously, then alternating 15-30 second images of each ureter or ureteral orifice will be obtained. The surgeon should note the time blue color is visualized in each ureter jet stream.

Blood samples for PK analysis Urine samples will be collected at 0-30 minutes and 30 minutes- 2 hours post Bludigo® injection.

All treated patients will have a follow-up visit 14 (± 3) days after the procedure. A final telephone call to assess adverse events (AEs) will occur at Day 30 (±2 days).

Safety assessments will include monitoring of vital signs, AEs and laboratory testing post the procedure.

DETAILED DESCRIPTION:
The study will enroll approximately 18 pediatric patients from approximately 2-3 study centers in the United States.

Patients scheduled for urological or gynecological surgical procedures who are < 17 years will be screened for participation.

A minimum of 6 patients will be enrolled in each of the following three age groups: birth to <6-years old, 6 to < 12 years old, 12 to < 17 years old.

Screening will occur within 30 days before study drug administration (Day of Surgery).

After signing the informed consent, review of inclusion and exclusion criteria will be performed. The collection of medical history and concomitant medications, the completion of a physical examination including vital signs measurement, ECG, and the collection of baseline laboratory testing (samples must be collected within 14 days of day 1) will be completed during the screening period.

On the Day of Surgery (Day 1) patients will be evaluated for eligibility for treatment.

To evaluate the efficacy outcomes, each patient will be injected with a weight-based dose of Bludigo® (0.05 mL/kg rounded up (if necessary) to a minimum of 0.5 mL) the maximum dose to be injected is not to exceed 2.5 mL. The ureteral orifices / urine jet will be observed, and a video will be recorded for 10 minutes. The time that will be captured on video is from the time of Bludigo® injection to 10 minutes post injection. If both ureters cannot be visualized simultaneously, then alternating 15-30 second images of each ureter or ureteral orifice will be obtained. The surgeon should note the time blue color is visualized in each ureter jet stream.

Blood samples for PK analysis Urine samples will be collected at 0-30 minutes and 30 minutes- 2 hours post Bludigo® injection.

All treated patients will have a follow-up visit 14 (± 3) days after the procedure. A final telephone call to assess adverse events (AEs) will occur at Day 30 (±2 days).

Safety assessments will include monitoring of vital signs, AEs and laboratory testing post the procedure.

ELIGIBILITY:
Inclusion Criteria:

I01. Patients from birth to < 17 years

I02. Patients whose Parents or Legal Authorized Representative (LAR) have signed a written, IRB approved, informed consent form (ICF) and applicable assent obtained.

I03. Patients scheduled for urological or gynecological surgical procedures in which the patency of the ureters must be assessed by the surgeon during the surgery.

Exclusion Criteria:

E01. For patients ≥ 1 year of age, Stage 5 Chronic Kidney Failure (defined as an eGFR (estimated glomerular filtration rate) ≤ 15mL/min/1.73 m2). (Calculated using the revised "Bedside Schwartz" equation (Schwartz et al. 2009) ). The revised "Bedside Schwartz" for eGFR is calculated as follows. eGFR (mL/min/1.73m2) = 0.413 * height/Scr, where height is baseline height measured in cm and Scr is baseline serum creatine measured in mg/dL;

For patients less than 1 year of age, measured serum creatinine greater than 1.5-times the upper limit of normal (>97.5 percentile) based on the reference table in Boer et al., 2010.

E02. Patients weighing less than 5 kgs.

E03. Patients with known severe hypersensitivity reactions to Bludigo® or other dyes including contrast agents.

E04. Patients with a history of, or being evaluated or treated for, gynecologic, renal, or urogenital (ureteral or bladder) cancer.

E05. Patients with known congenital cardiac conditions or who have a history of arrythmia, hypotension, hypertension, bradycardia or tachycardia.

E06. Patients, as assessed by the Investigator, with other conditions / concomitant diseases precluding their safe participation in this study (e.g., major systemic diseases).

E07. Unable to meet specific protocol requirements (e.g., scheduled visits), or has a condition that could lead to non-compliance with the study procedures or patient/parent/LAR uncooperative.

E08. Patient is the child of Investigator or any Sub-Investigator, research assistant, pharmacist, study coordinator, other staff or relative thereof directly involved in the conduct of the protocol.

E09. Patients with a life expectancy ≤ 6 months.

E10. Requirement for concomitant treatment with renal tubule transport inhibitors or with any treatment that could potentially discolor urine (see section 6.6)

E11. Patients who are pregnant or breast feeding.

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 18 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Responders to Bludigo® | 10 minutes post study drug administration
  Urine jet conspicuity scores based on the 5-point conspicuity score utilized in study PVP-19IC01 in adults. The 5-point scale is defined as:
  1. No jet observed
  2. Weak jet, little color contrast
  3. Color contrast or significant jet flow
  4. Strong jet flow with good color contrast
  5. Strong jet flow with striking contrast in color

SECONDARY OUTCOMES:
Time to visualization | 10 minutes post drug administration
  Time to visualization of blue color at each ureteral orifice following administration of Bludigo®.
Pharmacokinetics parameters | 2 hours post study drug administration
  Amount of Bludigo® excreted in urine.
Area under the curve | 40 minutes post study drug administration
  Area under the curve
Maximum plasma concentration (C max) | 40 minutes post study drug administration
  Maximum plasma concentration (C max)
Time to reach maximum plasma concentration (T max) | 40 minutes post study drug administration
  Time to reach maximum plasma concentration (T max)

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Boytim, Ph.D., Study Director — Provepharm SAS

IPD SHARING:
Plan to Share IPD: No